CLINICAL TRIAL: NCT01489618
Title: Randomised, Multicentric, Phase ii Study of the Immunogenicity of a "Prime Boost" Vaccination Strategy Combining Conjugated Anti- Pneumococcal Vaccine (s0) and Polysaccharide Anti- Pneumococcal Vaccine (s4) Compared to Polysaccharide Anti- Pneumococcal Vaccine Alone (s4) In Patients With Common Variable Immunodeficiency
Brief Title: "Prime Boost" Vaccination Strategy Combining Conjugated Anti- Pneumococcal Vaccine (s0) and Polysaccharide Anti- Pneumococcal Vaccine (s4) Compared to Polysaccharide Anti- Pneumococcal Vaccine Alone (s4) In Patients With Common Variable Immunodeficiency
Acronym: EVAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: End of production
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RBM04-34; 2007-003235-23 (EudraCT Number)
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Common Variable Immunodeficiency
Keywords: Common variable immunodeficiency; pneumococcal vaccine; prime boost
MeSH Terms: conditions — Common Variable Immunodeficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPS (Active Comparator): Group 1: patients will a single administration of the PPS (one dose at W4). 25 patients will be randomised in this group.
  Interventions: Biological: PPS
- PnCJ PPS (Experimental): Group 2: patients will receive a first boost with the PnCj (one dose at W0) and then one administration of the PPS vaccines (one dose at W4). 47 patients will be randomised in this group.
  Interventions: Biological: PnCJ PPS

INTERVENTIONS:
Biological: PPS — POLYSACCHARIDE ANTI- PNEUMOCOCCAL VACCINE
  Arms: PPS
Biological: PnCJ PPS — PRIMEBOOST CONJUGATED ANTI- PNEUMOCOCCAL VACCINE (Week 0) POLYSACCHARIDE ANTI- PNEUMOCOCCAL VACCINE (Week 4)
  Arms: PnCJ PPS

SUMMARY:
The main objective of this study is to evaluate and to compare the specific antibody response to a " prime-boost " vaccine strategy combining the seven valence pneumococcal conjugate vaccine (PnCj) prime at W0 followed by the administration of the pneumococcal capsular polysaccharide vaccine (PPS) boost at W4, to the administration of the pneumococcal capsular polysaccharide vaccine (PPS) alone at W4 in patients with common variable immunodeficiency.

DETAILED DESCRIPTION:
Main objective :

The main objective of this study is to evaluate and to compare the specific antibody response to a " prime-boost " vaccine strategy combining the seven valence pneumococcal conjugate vaccine (PnCj) prime at W0 followed by the administration of the pneumococcal capsular polysaccharide vaccine (PPS) boost at W4, to the administration of the pneumococcal capsular polysaccharide vaccine (PPS) alone at W4 in patients with common variable immunodeficiency.

Secondary objectives :

* Evaluation and comparison the specific antibody response to seven pneumococcal serotypes, shared by the PnCj and PPS vaccines (4, 6B, 9V, 14, 18C, 19F, 23F), and two serotypes of the PPS vaccine (1, 5) 4 weeks after the single (W8 for patients from Group 1) or the first vaccination (W4 for patients from group 2).
* Evaluation of the duration of the specific antibody response at week 24
* Evaluation of the T CD4 lymphocyte response (proliferation and cytokine production) to the CRM protein
* Study of the Immunoglobulin V gene repertoire (immunoscope) before and after vaccination.
* Safety of the vaccines
* Effect of the vaccine strategies on the frequency of Streptococcus pneumoniae infections (bronchitis, sinusitis and recurrent upper respiratory tract)

EXPERIMENTAL METHODS

Study design

Randomised, multicentric, controlled phase II study of the immunological efficacy of a "prime boost" strategy combining the sequential administration of the PnjC and PPS anti-pneumococcal vaccines, compared to the administration of the PPS vaccine alone, in patients with common variable immunodeficiency.

After randomisation (at W-4) 72 patients will be assigned to the two following groups:

* Group 1: patients will a single administration of the PPS (one dose at W4). 25 patients will be randomised in this group.
* Group 2: patients will receive a first boost with the PnCj (one dose at W0) and then one administration of the PPS vaccines (one dose at W4). 47 patients will be randomised in this group.

R : 1 :2 (Group1 :2)

The final evaluation of this study is at week 12; i.e 4 weeks after the administration of the PPS vaccine in the two groups of patients. A follow up of patients until week 48 will be proposed to patients in order to evaluate the duration of the antibody response at wek 48.

DURATION OF THE STUDY

* Inclusion period : 18 months
* vaccination period: 2 months
* Patients follow-up : 7 months

Number of patients : 72

PRIMARY AND SECONDARY EFFICACY ENDPOINTS

The pneumococcal conjugate vaccine (PnCj) vaccin contains the following 7 pneumococcal serotypes: 4, 6B, 9V, 14, 18C, 19F, 23F.

The pneumococcal capsular polysaccharide vaccine (PPS) contains 23 pneumococcal serotypes and shares the seven serotypes included in PnCJ.

Primary endpoint :

The primary end point of this study is the proportion of responders to each serotype contained in the PnjC vaccine in the two groups of this study according to 4 categories: 5-7; 3-4; 2-1 and 0. A responder is defined by a rise (at least two fold from baseline) of antibody titers specific to pneumococcal serotypes.

Secondary endpoints :

* The following parameters will be evaluated and compared in the two groups of the study : La réponse immunitaire anticorps vis-à-vis des différents sérotypes vaccinaux communs

  * geometric mean of the specific antibody titers
  * proportion of patients who experienced an increase of specific antibody levels >1 µg/ml
* Evaluation of the priming effect of the PnCj vaccine in the group 2
* Duration of the specific antibody reponses at week 24
* CD4 T lymphocyte responses to the CRM protein (proliferative and cytokine production) in the two groups of the study at weeks 0, 8 and 12.
* Safety of the vaccines
* Effect of the vaccine stategies on the frequency of Streptococcus pneumoniae infections (bronchitis, sinusitis and recurrent upper respiratory tract)

STATISTICAL CONSIDERATIONS

The initial hypothesis for this study is the superiority of the priming strategy. Expected responses are : 0% in group 1 (PPS alone) and 30% in group 2 (PnCj vace and PPS). The number of patients is based on power of 84%.

The primary end point is the proportion of responders to each serotype contained in the PnCj vaccine in the 2 groups. The percentage of patients in each group will be compared by a Fisher's exact test. Mann-Whitney test and Wilcoxon paired test will be used for the comparison of antibody levels and percentage of responding patients respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 65 years
* Common variable immunodeficiency according to the WHO criteria,
* Patients treated with intravenous or subcutaneous immunoglobulin.
* Written informed consent
* Absence of acute infections, or other evolutive diseases related to the (cancer, auto-immune disease…)

Exclusion Criteria:

* IgG subclass deficiency
* IgA selective deficiency,
* Other primary humoral deficiency (X-linked agammaglobulinemia, Hyper IgM syndrome),
* Long course treatment with corticosteroids > 5mg per day
* Chemotherapy in the last 3 years,
* Prior pneumococcal vaccination in the last 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
proportion of responders to each serotype | 8 weeks
  The primary end point of this study is the proportion of responders to each serotype contained in the PnjC vaccine in the two groups of this study according to 4 categories: 5-7; 3-4; 2-1 and 0. A responder is defined by a rise (at least two fold from baseline) of antibody titers specific to pneumococcal serotypes.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Immunologie Clinique Hôpital Henri Mondor, Créteil, France